CLINICAL TRIAL: NCT00873886
Title: A Study of the Pharmacology of Oseltamivir (Tamiflu) in Pregnancy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We will focus on other Tamiflu research studies. No subjects were enrolled.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Richard Beigi, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #PRO07080362; 5U10HD047905-02 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oseltamivir (Tamiflu) (Experimental)
  Interventions: Drug: Oseltamivir (Tamiflu)
- Esterase (Other)
  Interventions: Procedure: Blood Draws

INTERVENTIONS:
Drug: Oseltamivir (Tamiflu) — The following procedures will be performed on two occasions: once at least three days prior to the scheduled pregnancy termination procedure and again about eight weeks after the termination procedure.
  A) Subject will take 75 mg of oseltamivir pill by mouth
  B) Multiple blood draws (1 teaspoon each) over the next 48 hours after taking oseltamivir. Urine samples also will be collected.
  Arms: Oseltamivir (Tamiflu)
Procedure: Blood Draws — Two blood draws (1 teaspoon each) will be performed: once during third trimester of pregnancy and again about eight weeks after delivery.
  Arms: Esterase

SUMMARY:
The primary research question of this study is: Does the pharmacokinetics of oseltamivir after a single oral dose differ between the pregnant and non-pregnant women?

DETAILED DESCRIPTION:
With the pending threat of pandemic avian influenza, the disproportionate morbidity and mortality documented in previous 20th century pandemics among pregnant women, and the lack of any data for use of these vital antiviral drugs in pregnancy, study of the pharmacology of oseltamivir in pregnancy is imperative. If and when the next pandemic occurs, a better understanding of this drug's safety and pharmacologic profiles for use in pregnancy is critical given the fact that it will be used in this vulnerable patient population.

This is a pilot study of the use of oseltamivir in pregnancy. This data will be combined with data from the parallel Pediatric Pharmacology Research Unit (PPRU) studies to put together a portfolio for use in understudied populations. This will allow for a re-thinking of the current status and potentially allow for small trials to be performed with patients who are suffering from influenza in pregnancy, to assess efficacy. The relevance with the pandemic strain and its corresponding Minimum Inhibitory Concentration (MIC) may have direct implications for dosing in pregnancy if lower levels of drug are documented. In addition, depending on the findings from the esterase component of the investigation, future investigation into mechanistic bases for changes in enzyme activity are possible.

ELIGIBILITY:
Inclusion Criteria:

* For Oseltamivir (Tamiflu) arm:
* Singleton gestation prior to 24 0/7 weeks gestation
* Planning to undergo a termination procedure for the incident pregnancy
* Willingness to take the single-dose medication and to follow study procedures
* Able to undergo informed consent.
* For Esterase arm:
* Singleton gestation greater than 32 completed weeks and less than 40 completed weeks of gestation
* Absence of severe pregnancy complication that could affect body volume and or metabolism (i.e., preeclampsia, renal dysfunction, hepatic dysfunction [defined as serum creatinine clearance of < 30 ml/min or a known ALT/AST> 2x facility normal value], etc.)
* Willingness to follow study procedures
* Able to undergo informed consent
* The use of medications that may affect renal metabolism is not a contraindication to participation since these subjects are only undergoing PK sampling.

Exclusion Criteria:

* For Oseltamivir (Tamiflu) arm:
* Known current in utero fetal death
* Significant medical history and/or medication use as determined by the investigator that has the potential to affect results of the study or put the patient at risk from the single-dosing
* Known hypersensitivity to the components of the study drug
* Known hepatic or renal dysfunction (defined as serum creatinine clearance of < 30 ml/min or a known ALT/AST> 2x facility normal value)
* Chronic use of street drugs (obtained via subject interview and/or medical history)
* Participation in any other concurrent interventional study.
* We will ask if they have a history of depression in the past requiring treatment or if they are currently actively depressed. If either of these questions yields a positive response, we will not consider the patient eligible and will not enroll the subject.
* For Esterase arm:
* Known current in utero fetal death
* Significant medical history as determined by the investigator to potentially affect results of the study
* Chronic use of street drugs (obtained via subject interview and/or medical history
* Participation in any other concurrent interventional study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Change in the area under the concentration vs. time curve (AUC 0-7 d) in the first and second trimesters of pregnancy with comparisons to the post-termination non-pregnant follow-up data on these enrollees and historical non-pregnant data. | Less than 9 weeks for subjects planning termination; up to 5 months for subjects enrolled during their 3rd trimester.

SECONDARY OUTCOMES:
Non-compartmental model analysis for Cmax, Tmax, Cl/F, Clr,V/F, MRT and t ½. | Less than 9 weeks for subjects planning termination; up to 5 months for subjects enrolled during their 3rd trimester.
Plasma concentrations of oseltamivir after single-dosing. | Less than 9 weeks for subjects planning termination; up to 5 months for subjects enrolled during their 3rd trimester.
Evaluation of carboxy-esterase levels and activity in all trimesters of pregnancy with comparison to the post-partum internal controls. | Less than 9 weeks for subjects planning termination; up to 5 months for subjects enrolled during their 3rd trimester.
Tolerance (side effect profile) of single-dose oseltamivir in pregnancy. | Less than 9 weeks for subjects planning termination; up to 5 months for subjects enrolled during their 3rd trimester.

CONTACTS AND LOCATIONS:
Overall Officials: Richard H. Beigi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Advisory Committee on Immunization Practices; Smith NM, Bresee JS, Shay DK, Uyeki TM, Cox NJ, Strikas RA. Prevention and Control of Influenza: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2006 Jul 28;55(RR-10):1-42. PMID 16874296
- [Background] Neuzil KM, Reed GW, Mitchel EF, Simonsen L, Griffin MR. Impact of influenza on acute cardiopulmonary hospitalizations in pregnant women. Am J Epidemiol. 1998 Dec 1;148(11):1094-102. doi: 10.1093/oxfordjournals.aje.a009587. PMID 9850132
- [Background] Irving WL, James DK, Stephenson T, Laing P, Jameson C, Oxford JS, Chakraverty P, Brown DW, Boon AC, Zambon MC. Influenza virus infection in the second and third trimesters of pregnancy: a clinical and seroepidemiological study. BJOG. 2000 Oct;107(10):1282-9. doi: 10.1111/j.1471-0528.2000.tb11621.x. PMID 11028582
- [Background] Cox S, Posner SF, McPheeters M, Jamieson DJ, Kourtis AP, Meikle S. Hospitalizations with respiratory illness among pregnant women during influenza season. Obstet Gynecol. 2006 Jun;107(6):1315-22. doi: 10.1097/01.AOG.0000218702.92005.bb. PMID 16738158
- [Background] Cox S, Posner SF, McPheeters M, Jamieson DJ, Kourtis AP, Meikle S. Influenza and pregnant women: hospitalization burden, United States, 1998-2002. J Womens Health (Larchmt). 2006 Oct;15(8):891-3. doi: 10.1089/jwh.2006.15.891. PMID 17087611
- [Background] Lindsay L, Jackson LA, Savitz DA, Weber DJ, Koch GG, Kong L, Guess HA. Community influenza activity and risk of acute influenza-like illness episodes among healthy unvaccinated pregnant and postpartum women. Am J Epidemiol. 2006 May 1;163(9):838-48. doi: 10.1093/aje/kwj095. Epub 2006 Mar 22. PMID 16554352
- [Background] ACOG Committee on Obstetric Practice. ACOG committee opinion number 305, November 2004. Influenza vaccination and treatment during pregnancy. Obstet Gynecol. 2004 Nov;104(5 Pt 1):1125-6. PMID 15516422
- [Background] Garcia-Sastre A, Whitley RJ. Lessons learned from reconstructing the 1918 influenza pandemic. J Infect Dis. 2006 Nov 1;194 Suppl 2:S127-32. doi: 10.1086/507546. PMID 17163385
- [Background] Webster RG, Govorkova EA. H5N1 influenza--continuing evolution and spread. N Engl J Med. 2006 Nov 23;355(21):2174-7. doi: 10.1056/NEJMp068205. No abstract available. PMID 17124014
- [Background] Ferguson NM, Cummings DA, Cauchemez S, Fraser C, Riley S, Meeyai A, Iamsirithaworn S, Burke DS. Strategies for containing an emerging influenza pandemic in Southeast Asia. Nature. 2005 Sep 8;437(7056):209-14. doi: 10.1038/nature04017. Epub 2005 Aug 3. PMID 16079797
- [Background] Moscona A. Neuraminidase inhibitors for influenza. N Engl J Med. 2005 Sep 29;353(13):1363-73. doi: 10.1056/NEJMra050740. No abstract available. PMID 16192481
- [Background] Dutkowski R, Thakrar B, Froehlich E, Suter P, Oo C, Ward P. Safety and pharmacology of oseltamivir in clinical use. Drug Saf. 2003;26(11):787-801. doi: 10.2165/00002018-200326110-00004. PMID 12908848
- [Background] Health Sciences Authority. Product Safety Alert: new preclinical findings on Oseltamivir. March 2004. (Accessed November 27, 2006 at: http://www.hsa.gov.sg/docs/safetyalert_oseltamivir_March04.pdf.)
- [Background] Hayden FG, Treanor JJ, Betts RF, Lobo M, Esinhart JD, Hussey EK. Safety and efficacy of the neuraminidase inhibitor GG167 in experimental human influenza. JAMA. 1996 Jan 24-31;275(4):295-9. PMID 8544269
- [Background] Massarella JW, He GZ, Dorr A, Nieforth K, Ward P, Brown A. The pharmacokinetics and tolerability of the oral neuraminidase inhibitor oseltamivir (Ro 64-0796/GS4104) in healthy adult and elderly volunteers. J Clin Pharmacol. 2000 Aug;40(8):836-43. doi: 10.1177/00912700022009567. PMID 10934667
- [Background] Ward P, Small I, Smith J, Suter P, Dutkowski R. Oseltamivir (Tamiflu) and its potential for use in the event of an influenza pandemic. J Antimicrob Chemother. 2005 Feb;55 Suppl 1:i5-i21. doi: 10.1093/jac/dki018. PMID 15709056